CLINICAL TRIAL: NCT07387926
Title: Open-label, Phase I/II Study to Evaluate Safety and Efficacy of Asciminib With Chemotherapy Followed by Asciminib Plus Blinatumomab in Pediatric, Adolescent, and Young Adults With Relapsed or Refractory BCR::ABL1-positive (Philadelphia Positive, Ph+) or BCR::ABL1-like (Ph-like) ALL
Brief Title: Safety and Efficacy of Asciminib in Pediatrics and Young Adults With Relapse/Refractory (r/r) Philadelphia Positive (Ph+) or ABL-class Ph-like Acute Lymphoblastic Leukemia (ALL)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001L12101; 2025-522019-40 (EudraCT Number)
Record Dates: First submitted 2026-01-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive; Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Keywords: Asciminib; ABL001; Ph+ chromosome acute lymphoblastic leukemia; ABL1/ABL2 fusion Ph-like ALL; BCR::ABL1; blinatumomab; dexamethasone; vincristine; chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asciminib; Dexamethasone; Vincristine; blinatumomab; Methotrexate; Cytarabine; Hydrocortisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Asciminib Adult formulation group: escalating doses evaluated
  Asciminib Pediatric formulation group: dose is based on body weight; dose level being evaluated will be converted into a mg/kg daily dose.
  Interventions: Drug: Asciminib Adult formulation; Drug: Asciminib Pediatric formulation; Drug: Dexamethasone; Drug: Vincristine; Drug: Blinatumomab; Drug: Methotrexate (intrathecal); Drug: Cytarabine (intrathecal); Drug: Hydrocortisone (intrathecal); Drug: Prednisolone (intrathecal)

INTERVENTIONS:
Drug: Asciminib Adult formulation — oral, administered daily; Cycles 1, 2, 3
  Other Names: ABL001
Drug: Asciminib Pediatric formulation — oral, administered daily; Cycles 1, 2, 3
  Other Names: ABL001
Drug: Dexamethasone — Fixed doses, oral (preferred) or intravenous (IV) twice daily; Cycle 1, Days 1 - 14; (Cycle 1 = 28 days)
Drug: Vincristine — Fixed doses, IV, weekly; Cycle 1
Drug: Blinatumomab — Dosing based on bone marrow disease burden and weight. Continuous IV infusion; Cycles 2, 3
Drug: Methotrexate (intrathecal) — Intrathecal
Drug: Cytarabine (intrathecal) — Intrathecal
Drug: Hydrocortisone (intrathecal) — Intrathecal
Drug: Prednisolone (intrathecal) — Intrathecal

SUMMARY:
Multi-center, open-label, single arm study of asciminib in participants aged ≥1 year to ≤30 years old with r/r Ph+ or ABL-class Ph-like ALL. This study will have 2 parts: Part 1 dose escalation and Part 2 dose expansion. Part 1 dose escalation will enroll participants aged ≥1 year to ≤30 years to determine the recommended phase 2 dose (RP2D) of asciminib when administered with low intensity chemotherapy. Part 2 dose expansion will enroll participants aged ≥1 year to ≤30 years to evaluate safety, tolerability, and efficacy of asciminib at the RP2D with the treatment regimen.

DETAILED DESCRIPTION:
This is a single arm phase I/II multicenter study to assess the safety and efficacy of asciminib at the RP2D in combination with low intensity chemotherapy (debulking induction) followed by asciminib plus blinatumomab (consolidation) in pediatric and young adult participants with r/r Ph+ ALL (inclusive of participants with T315I mutation).

A separate cohort on this study will enroll participants with r/r ABL-class Ph-like ALL (inclusive of participants with T315I mutation).

The aim of the study design is to explore a novel treatment regimen which is expected to be more tolerable than the high intensity chemotherapy backbone-based regimens.

This study will consist of a 2-part design:

1. Part 1 dose escalation using a Bayesian Optimal Interval (BOIN) statistical design, and after determination of RP2D,
2. Part 2 dose expansion

Participants will only enroll in either Part 1 or Part 2, and not both.

Both Part 1 and Part 2 (dose escalation and dose expansion) will have the following phases:

* Core Study Treatment Phase
* Survival Follow up Phase

The core study treatment phase will consist of 3 cycles of therapy: cycle 1 asciminib with low intensity chemotherapy (debulking induction), followed by cycle 2 (blinatumomab-block 1 with asciminib) and cycle 3 (blinatumomab-block 2 with asciminib).

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Ph+ ALL or ABL1 or ABL2 fusion Ph-like ALL, inclusive of participants with ABL1 T315I mutations
* Participants with CNS1, CNS2, CNS3a, or CNS3b at screening
* Active B-Cell ALL at screening defined by MFC or IG/TCR PCR of ALL blasts >0.01% in participants with either:

  1. Primary refractory disease (>0.01% ALL blasts present at the end of consolidation) OR
  2. Relapsed ALL with evidence of involvement of BM with ALL (MFC or IG/TCR PCR >0.01%) after at least one line of therapy
* Documented history of CD19 expressing B-cell ALL (in peripheral blood or bone marrow by flow cytometry).

  a) For participants who received anti-CD19 targeted therapy (e.g CD19 CAR T cells or blinatumomab), CD19 expressing B-cell ALL must be documented after anti-CD19 therapy completion prior to cycle 1 day 1
* Adequate hepatic and renal function (local laboratory analysis) as defined:

  1. ALT ≤ 5x upper limit of normal (ULN) for age
  2. Total bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x ULN) for age, except for participants with Gilbert's syndrome who may only be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
  3. Estimated glomerular filtration rate (eGFR) using the Cockcroft-Gault formula in participants ≥ 18 years, OR radioisotope GFR ≥50 mL/min/1.73 m^2, OR creatinine based on age and sex for participants < 18 years old
* Adequate cardiac function defined as shortening fraction ≥27% by echocardiogram (ECHO) OR left ventricular ejection fraction of ≥50% by ECHO

Exclusion Criteria:

* Participants with >3 relapses of ALL
* Extramedullary disease (non-CNS and/or isolated CNS disease)
* Participants with CNS3c (Clinical signs of CNS leukemia (such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome))
* Cardiac or cardiac repolarization abnormality, including but not limited to clinically significant cardiac arrhythmias, long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or other clinically significant heart disease (e.g., congestive heart failure, etc.)
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-26 (Estimated); Primary Completion 2033-01-10 (Estimated); Study Completion 2035-12-12 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Escalation: To determine the Recommended Phase II Dose (RP2D) of asciminib when administered with low intensity chemotherapy | During Cycle 1 (Cycle 1 = 28 days)
  An integrated assessment of tolerability, safety profiles, dose-limiting toxicities (DLTs), treatment responses, and available pharmacokinetic (PK) data.
Part 2 Dose Expansion: Assess the rate of complete remission (CR) at RP2D | End of Cycle 1 (Cycle 1 = 28 days)
  Percentage of participants achieving complete remission (CR)

SECONDARY OUTCOMES:
Complete remission (CR) rate | End of Cycle 2 and Cycle 3 (Cycle 2 & 3 = 42 days)
  Percentage of participants achieving CR
Overall response rate (ORR) | At and by the end of Cycle 1 (Cycle 1 = 28 days), Cycle 2, and Cycle 3 (Cycle 2 & 3 = 42 days)
  Percentage of participants who had CR and/or complete remission with incomplete blood count recovery (CRi)
Next generation sequencing (NGS) minimal residual disease (MRD) negative rate | At and by the end of Cycle 1 (Cycle 1 = 28 days), Cycle 2, and Cycle 3 (Cycle 2 & 3 = 42 days)
  Percentage of participants achieving NGS MRD negative CR/CRi
Multiparametric flow cytometry (MFC) MRD negative CR/CRi rate | At and by the end of Cycle 1 (Cycle 1 = 28 days), Cycle 2, and Cycle 3 (Cycle 2 & 3 = 42 days)
  Percentage of participants achieving MRD negative CR/CRi
Disease Free Survival (DFS) | End of Cycle 3 (Cycle 3 = 42 days) in Part 2 of the study and at the end of study (EOS = approx. 3 years)
  The period from when a participant is in remission until they have relapse or death due to any reason.
Overall survival (OS) | End of Cycle 3 (Cycle 3 = 42 days) in Part 2 of the study and at the end of study (EOS = approx. 3 years)
  The duration of time from treatment initiation until the participant's death due to any reason.
Pharmacokinetic (PK) parameter of asciminib at steady state: AUClast | Cycle 1, Day 8 (Cycle 1 = 28 days)
  Area Under the Curve to the Last Measurable Concentration-represents the total drug exposure (area under the plasma concentration-time curve) from the time of administration until the last measurable concentration
PK parameter of asciminib at steady state: Cmax | Cycle 1, Day 8 (Cycle 1 = 28 days)
  Maximum concentration-the peak (highest) plasma drug concentration observed after administration
PK parameter of asciminib at steady state: Tmax | Cycle 1, Day 8 (Cycle 1 = 28 days)
  The time it takes to reach the Cmax after drug administration
PK parameter of asciminib at steady state: Ctrough | Cycle 1, Day 8 (Cycle 1 = 28 days); Cycle 2, Day 22 (Cycle 2 = 42 days); Cycle 3, Day 22 (Cycle 3 = 42 days)
  Trough concentration- lowest drug concentration observed, typically right before the next dose is administered (steady-state condition)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
Supporting Information: Study Protocol
URL: https://www.clinicalstudydatarequest.com